CLINICAL TRIAL: NCT02618551
Title: Evaluation of the Efficiency of Bronchial Thermoplasty on Dynamic Hyperinflation in Uncontrolled Severe Asthma
Brief Title: Bronchial Thermoplasty for Severe Asthma With Dynamic Hyperinflation
Acronym: HEAT-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/14/7422
Record Dates: First submitted 2015-11-26; First posted 2015-12-01 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Asthma; Hyperinflation
Keywords: Thermoplasty; Severe asthma; Dynamic hyperinflation
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Patients will be treated by three bronchial thermoplasty sessions.
  Interventions: Procedure: Bronchial thermoplasty for treatment of severe asthma

INTERVENTIONS:
Procedure: Bronchial thermoplasty for treatment of severe asthma — Three sessions of bronchial thermoplasty are needed to treat patients. There will be 3 to 4 weeks between each procedure.
  Bronchial thermoplasty procedure is performed under general anesthesia. The medical device used in this research to achieve the thermoplasty is the Alair system (class IIb medical device ; Boston scientific)
  A confocal endomicroscopy will be conducted at the first and final session of thermoplasty. This examination involves analyzing and recording the structure of bronchi microscopy through a small catheter placed on the bronchus. Photographs of the bronchi will be realized.

SUMMARY:
Bronchial thermoplasty is a treatment for severe asthma that consist in decreasing the thickness of bronchial muscle by heat using a catheter inserted into the bronchi under direct vision with the help of an endoscope This treatment has shown efficacy on symptoms, quality of life and the number of exacerbations related to severe asthma.

This clinical study evaluates the efficiency of this treatment on the dynamic hyperinflation phenomenon (worsening of bronchial obstruction during exercise in patients with asthma contributing to worsening shortness of breath).

DETAILED DESCRIPTION:
Bronchial thermoplasty is a recently validated bronchoscopic technique for the management of severe asthma that treats smooth muscle by radiofrequency to reduce its thickness. This procedure leads to improved asthma control and quality of life, but also to decreased exacerbations frequency and number of emergencies hospitalizations. This treatment requires 3 procedures every 3 to 4 weeks.

The pathophysiological mechanisms underlying its effectiveness need to be better understood for an improved selection of best candidates. In particular, there is a discrepancy between the improvement observed in symptoms (ACQ), quality of life (AQLQ) and the lack of improvement in forced expiratory volume in 1 second (FEV1). Investigator assume that this paradox is due to an efficiency appearing at effort, targeting dynamic hyperinflation phenomenon.

The objective of this study is to evaluate the influence of bronchial thermoplasty on dynamic hyperinflation in severe asthma. The secondary objectives are to assess the effectiveness of bronchial thermoplasty (ACQ, AQLQ) in a selected population of patients with dynamic hyperinflation and to describe bronchial wall structural changes by probe-based confocal LASER endomicroscopy (pCLE).

ELIGIBILITY:
Inclusion Criteria:

* Severe asthma, uncontrolled despite optimal treatment according to GINA (global initiative for asthma) recommendations
* At least 2 exacerbations treated by systemic steroids in the last year
* FEV1 between 40 and 80% of predicted values and dynamic hyperinflation (defined as a decrease in inspiratory capacity by more than 500 ml during exercise)

Exclusion Criteria:

* Current asthma exacerbation or respiratory infection
* History of exacerbation after bronchoscopy
* FEV1 < 40% of predicted values
* Oxygen saturation < 90%
* Contra-indications to ALAIR catheter system : pacemaker or other electronic implanted device
* Allergy to Remifentanyl or Propofol
* pregnancy; breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Evolution of dynamic hyperinflation | 3 months
  A lung plethysmography will be used to patients to see evolution of dynamic hyperinflation after bronchial thermoplasty, defined as a decrease in inspiratory capacity by more than 500 ml during exercise.
  The plethysmography will be made before the first procedure and three months after the third procedure.

SECONDARY OUTCOMES:
Structural modification of the bronchial wall | 3 months
  Description of structural modification of the bronchial wall by probe-based confocal LASER endomicroscopy (pCLE) induced by bronchial thermoplasty
Efficiency of bronchial thermoplasty on asthma | 3 months
  Efficiency of bronchial thermoplasty on asthma control (ACQ) and quality of life (AQLQ) in a selected population of patients with severe asthma with dynamic hyperinflation.
Assess side effects | 3 months
  Listing of thermoplasty complications (bronchitis, bronchospasm, exacerbation of asthma, hemoptysis, bronchiectasis) by medical staff

CONTACTS AND LOCATIONS:
Overall Officials: Alain DIDIER, MD, Principal Investigator — Toulouse Rangueil Larrey University Hospital
Locations (1):
- DIDIER Alain, Toulouse, Midi Pyrenees, France

REFERENCES:
- [Background] Moore WC, Bleecker ER, Curran-Everett D, Erzurum SC, Ameredes BT, Bacharier L, Calhoun WJ, Castro M, Chung KF, Clark MP, Dweik RA, Fitzpatrick AM, Gaston B, Hew M, Hussain I, Jarjour NN, Israel E, Levy BD, Murphy JR, Peters SP, Teague WG, Meyers DA, Busse WW, Wenzel SE; National Heart, Lung, Blood Institute's Severe Asthma Research Program. Characterization of the severe asthma phenotype by the National Heart, Lung, and Blood Institute's Severe Asthma Research Program. J Allergy Clin Immunol. 2007 Feb;119(2):405-13. doi: 10.1016/j.jaci.2006.11.639. PMID 17291857
- [Background] Brown RH, Wizeman W, Danek C, Mitzner W. Effect of bronchial thermoplasty on airway distensibility. Eur Respir J. 2005 Aug;26(2):277-82. doi: 10.1183/09031936.05.00006605. PMID 16055876
- [Background] Cox G, Thomson NC, Rubin AS, Niven RM, Corris PA, Siersted HC, Olivenstein R, Pavord ID, McCormack D, Chaudhuri R, Miller JD, Laviolette M; AIR Trial Study Group. Asthma control during the year after bronchial thermoplasty. N Engl J Med. 2007 Mar 29;356(13):1327-37. doi: 10.1056/NEJMoa064707. PMID 17392302
- [Background] Pavord ID, Cox G, Thomson NC, Rubin AS, Corris PA, Niven RM, Chung KF, Laviolette M; RISA Trial Study Group. Safety and efficacy of bronchial thermoplasty in symptomatic, severe asthma. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1185-91. doi: 10.1164/rccm.200704-571OC. Epub 2007 Sep 27. PMID 17901415
- [Background] Castro M, Rubin AS, Laviolette M, Fiterman J, De Andrade Lima M, Shah PL, Fiss E, Olivenstein R, Thomson NC, Niven RM, Pavord ID, Simoff M, Duhamel DR, McEvoy C, Barbers R, Ten Hacken NH, Wechsler ME, Holmes M, Phillips MJ, Erzurum S, Lunn W, Israel E, Jarjour N, Kraft M, Shargill NS, Quiring J, Berry SM, Cox G; AIR2 Trial Study Group. Effectiveness and safety of bronchial thermoplasty in the treatment of severe asthma: a multicenter, randomized, double-blind, sham-controlled clinical trial. Am J Respir Crit Care Med. 2010 Jan 15;181(2):116-24. doi: 10.1164/rccm.200903-0354OC. Epub 2009 Oct 8. PMID 19815809
- [Background] Wechsler ME, Laviolette M, Rubin AS, Fiterman J, Lapa e Silva JR, Shah PL, Fiss E, Olivenstein R, Thomson NC, Niven RM, Pavord ID, Simoff M, Hales JB, McEvoy C, Slebos DJ, Holmes M, Phillips MJ, Erzurum SC, Hanania NA, Sumino K, Kraft M, Cox G, Sterman DH, Hogarth K, Kline JN, Mansur AH, Louie BE, Leeds WM, Barbers RG, Austin JH, Shargill NS, Quiring J, Armstrong B, Castro M; Asthma Intervention Research 2 Trial Study Group. Bronchial thermoplasty: Long-term safety and effectiveness in patients with severe persistent asthma. J Allergy Clin Immunol. 2013 Dec;132(6):1295-302. doi: 10.1016/j.jaci.2013.08.009. Epub 2013 Aug 30. PMID 23998657
- [Derived] Guibert N, Guilleminault L, Lepage B, Heluain V, Fumat R, Dupuis M, Faviez G, Plat G, Hermant C, Didier A. Bronchial thermoplasty in patients with dynamic hyperinflation: results from the proof-of-concept HEAT trial. Eur Respir J. 2021 Jan 28;57(1):2001616. doi: 10.1183/13993003.01616-2020. Print 2021 Jan. No abstract available. PMID 32817006